CLINICAL TRIAL: NCT04577807
Title: Lerapolturev (Formerly Known as PVSRIPO) With or Without Immune Checkpoint Blockade in Advanced PD-1 Refractory Melanoma
Brief Title: LUMINOS-102: Lerapolturev With or Without Immune Checkpoint Blockade in Advanced PD-1 Refractory Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUMINOS-102
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Lerapolturev (Experimental): Lerapolturev (up to 1.6x10^9 TCID50) administered via direct injection of up to 6 lesions
  Interventions: Biological: Lerapolturev
- Arm 2: Lerapolturev and anti-PD-1 (Experimental): Lerapolturev (up to 1.6x10^9 TCID50) administered via direct injection of up to 6 lesions. Anti-PD-1 therapy given as per the anti-PD-1 approved package insert.
  Interventions: Biological: Lerapolturev; Biological: Anti-PD-1 Checkpoint Inhibitor

INTERVENTIONS:
Biological: Lerapolturev — Lerapolturev administered via direct lesion injection
Biological: Anti-PD-1 Checkpoint Inhibitor — Anti-PD-1 Checkpoint Inhibitor administered per package insert instructions
  Arms: Arm 2: Lerapolturev and anti-PD-1

SUMMARY:
A Phase 2 study to investigate the efficacy and safety of lerapolturev alone or in combination with a programmed death receptor-1 (anti-PD-1) inhibitor.

DETAILED DESCRIPTION:
This multi-center, open-label, randomized, Phase 2 will investigate the efficacy and safety of lerapolturev alone (Arm 1) or in combination with an anti-PD-1 inhibitor (Arm 2). Following a 6 participant safety run-in period, up to approximately 50 participants with cutaneous melanoma who previously failed anti-PD-1/L1-based therapy will be randomized 1:1 to receive either lerapolturev or lerapolturev plus an anti-PD-1.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Prior CDC-recommended vaccination series against PV, and has received a boost immunization with trivalent IPOL® (Sanofi-Pasteur SA) at least 1 week, but less than 6 weeks, prior to Day 1

   a. NOTE: Patients who are unsure of their vaccination status must provide evidence of anti-PV immunity prior to enrollment, as applicable
3. Has biopsy proven unresectable cutaneous melanoma and is willing to undergo tumor biopsy prior to the first dose of study drugs and at prespecified intervals during the study

   1. Patients with ocular, acral or mucosal melanoma are not eligible
   2. Patients with M1c or M1d disease are NOT eligble.
   3. Submission of an archival biopsy sample is allowed in lieu of the baseline tumor biopsy, provided the tissue is ≤4 months old and the participant received no intervening systemic/intratumoral anti-cancer therapy since the biopsy was acquired.
   4. Must have at least 1 lesion that is amenable to biopsy. The lesion must be safely accessible as determined by the investigator and should not be located at sites that require significant risk procedures to biopsy. Examples of sites considered to be of significant risk include but are not limited to the following: the brain, lung, mediastinum, pancreas, or endoscopic procedures extending beyond the esophagus, stomach, or bowel wall.
4. Has ≥ 2 melanoma lesions that are accurately measurable by caliper or a radiological method according to RECIST 1.1 criteria

   1. One lesion must be injectable- defined as a visible or palpable cutaneous, subcutaneous, or nodal melanoma lesion ≥10 mm in longest diameter or multiple injectable melanoma lesions which in aggregate have a longest diameter of ≥10 mm and where the minimum lesion size is ≥5 mm
   2. Note that visceral lesions (eg, liver, lung, retroperitoneal, subpleural lesions) are not considered injectable for the purposes of this trial.
5. Has had confirmed progression of disease (PD) while receiving at least 6 weeks (> 1 dose) of an FDA-approved anti-PD-1/L1 therapy (as monotherapy or in combination) for the treatment of melanoma. Note the following details:

   1. Initial PD as defined by RECIST v1.1
   2. Confirmation of PD per iRECIST must occur by repeat assessment ≥ 4 weeks from initial evidence of PD, in the absence of rapid clinical progression.
   3. Those who discontinue anti-PD-1/L1 therapy after at least 6 weeks (> 1 dose) and have confirmed PD per iRECIST within 12 weeks of their last anti-PD-1/L1 dose are also eligible, provided the anti-PD-1/L1 was not stopped due to toxicity requiring permanent discontinuation
   4. Those treated with anti-PD-1/L1 in the adjuvant setting and who have biopsy-confirmed progression either while receiving anti-PD-1/L1-based therapy or ≤ 12 weeks after their last dose of anti-PD-1/L1 therapy are allowed NOTE: Adjuvant is defined as therapy received after surgical resection of disease such that the patient has no evidence of disease when the anti-PD-1/L1 therapy is initiated. Patients with known BRAF mutation must have also failed or refused to receive BRAF-targeted therapy (alone or in combination with MEK inhibitor) to be eligible.
6. Eastern Cooperative Oncology Group (ECOG) status of 0-1
7. Serum lactate dehydrogenase (LDH) levels ≤ 3 x upper limit of normal (ULN)
8. Adequate bone marrow, liver and renal function as assessed by the following:

   1. Hemoglobin ≥ 9.0 g/dl, patients may be transfused
   2. Lymphocyte count ≥ 0.5 x 10^9/L (500 µL)
   3. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1500 µL)
   4. Platelet count ≥ 100 x 10^9/L (100,000 µL) without transfusion
   5. AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions: Patients with documented liver metastases: AST and ALT ≤ 5 x ULN; Patients with documented liver or bone metastases: ALP ≤ 5 x ULN
   6. Serum bilirubin ≤ 1.5 x ULN with the following exception: Patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN
   7. Measured or calculated (per institutional standards) creatinine clearance ≥ 30 ml/min (GRF can also be used in place of creatinine clearance)
   8. For patients not receiving therapeutic anticoagulation: INR, PT, PTT (or aPTT) ≤ 1.5 x ULN
9. Life expectancy of >12 weeks
10. Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for the study, and is willing/able to participate in the study

Exclusion Criteria:

1. Has biopsy-proven ocular, acral or mucosal melanoma
2. Has M1c or M1d disease
3. No more than one prior systemic anti-cancer regimen (monotherapy or combination) for management of melanoma. Additional details noted below:

   1. Adjuvant anti-cancer therapy administered ≥ 6 months prior to the first injection of lerapolturev does NOT count as a line of treatment.
   2. Patients with BRAF mutant melanoma may enroll if they have received ≤ 2 prior lines of systemic anti-cancer therapy only if one of those lines of therapy was a BRAF-targeted regimen (alone or in combination with MEK inhibitor).
   3. A line of therapy is defined as a regimen in which at least 2 doses of systemic anti-cancer therapy (monotherapy or combination) was administered, and the regimen was discontinued because of progressive disease
4. Uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry.

   1. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
   2. Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment
5. Grade ≥2 pleural effusion, pericardial effusion, or ascites
6. Active or history of autoimmune disease or immune deficiency within previous 2 years, with the following exceptions:

   1. History of autoimmune-related endocrinopathy (e.g. adrenal insufficiency, hypothyroidism, Type 1 diabetes mellitus, etc.) that is managed by hormone replacement therapy (e.g. hydrocortisone, thyroid hormone, insulin, etc.)
   2. Eczema, psoriasis, or lichen simplex chronicus with dermatologic manifestations only (eg, patients with psoriatic arthritis are excluded), provided all of the following conditions are met:

   i. Rash must cover <10% of body surface area

   ii. Disease is well-controlled at baseline and requires only low-potency topical corticosteroids

   iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within 12 months of Day 1
7. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

   a. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
8. History of a positive HIV RNA test (HIV 1 or 2 RNA by PCR)
9. Known active hepatitis B virus (HBV) infection (chronic or acute)

   a. NOTE: Participants with a negative HBsAg test and a positive total hepatitis B core antibody (HBcAb) test are allowed.
10. Known active hepatitis C virus (HCV) infection

    a. NOTE: History of a positive HCV antibody test, but negative HCV RNA test is allowed.
11. Active tuberculosis
12. Significant cardiovascular disease, such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months of Day 1, unstable arrhythmia, or unstable angina
13. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 elimination half-lives- whichever is shorter, prior to treatment, or has not recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy are eligible

    1. Note: Anti-PD-1/L1 within 4 weeks prior to Day 1 is allowed
    2. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
14. History of other malignancy within 2 years prior to Day 1, with the exception of those with a negligible risk of metastasis or death (e.g., resected cutaneous basal cell carcinoma, or other cancers with 5-year OS of >90%)
15. Severe infection within 4 weeks prior to Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia

    a. Prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are allowed.
16. Prior allogeneic stem cell or solid organ transplantation
17. Treatment with a live, attenuated vaccine within 4 weeks prior to Day 1
18. Treatment with systemic immunosuppressive medication within 4 weeks prior to Day 1, with the following exceptions:

    1. Participants who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible
    2. Patients receiving mineralocorticoids (e.g., fludrocortisone), or systemic prednisone equivalent corticosteroid doses of <10mg per day are eligible for the study
19. Known hypersensitivity to pembrolizumab, nivolumab, or any of the respective excipients
20. Requires therapeutic anticoagulation and cannot discontinue anticoagulation safely during the day prior, day of, and day after each lerapolturev injection

    a. NOTE: Participants receiving anticoagulation with warfarin at the time of study entry are allowed if they can be transitioned to an alternative anticoagulant (eg, low molecular weight heparin or direct oral anticoagulants) prior to the first dose of lerapolturev. Anyone transitioned from warfarin to an oral anticoagulant prior to the first dose of lerapolturev should have an INR <1.5x upper limit of normal in order to participate. Antiplatelet agents (eg, aspirin, clopidogrel, etc.) are not considered anticoagulants for the purposes of this study (ie, are allowed)
21. A pregnant or nursing female, or women of child-bearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception starting from signed ICF through 150 days after last anti-PD-1 dose
22. History of human serum albumin allergy
23. History of neurological complications due to polio virus infection
24. History of agammaglobulinemia
25. Concurrent participation in a separate interventional clinical trial during this study.
26. Any underlying medical condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromises the participant's well-being) or that could prevent, limit, or confound protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Orlando Health U7 Health Cancer Center, Orlando, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Treatment Centers of America, Zion, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Pittsburgh Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology -Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia University Medical Center, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety-run in: lerapolturev, up to 6x10^8 TCID50, administered on days 1, 10 and every 3 weeks thereafter. Total dose dependent on number and size of injectable lesions. Data are included in the Arm 1: lerapolturev Q3W group.
Groups:
- Arm 1: Lerapolturev QW: Lerapolturev, up to 1.6x10^9 TCID50, administered via direct injection. Weekly for 7 weeks and every 3 weeks thereafter.
  Total dose dependent on number and size of injectable lesions.
- Arm 1: Lerapolturev Q3W: Lerapolturev, up to 1.6x10^9 TCID50, administered every 3 weeks. Total dose dependent on number and size of injectable lesions.
- Arm 2: Lerapolturev and Anti-PD-1 QW: Lerapolturev, up to 1.6x10^9 TCID50, administered via direct injection. Weekly for 7 weeks and every 3 or 4 weeks thereafter.
  Total dose dependent on number and size of injectable lesions.
  Anti-PD-1 therapy given as per the anti-PD-1 approved package insert. Anti-PD-1 therapy was physician's choice of pembrolizumab or nivolumab.
- Arm 2: Lerapolturev and Anti-PD-1 Q3/Q4W: Lerapolturev, up to 1.6x10^9 TCID50, administered via direct injection every 3 or 4 weeks. Total dose dependent on number and size of injectable lesions.
  Anti-PD-1 therapy given as per the anti-PD-1 approved package insert. Anti-PD-1 therapy was physician's choice of pembrolizumab or nivolumab.
Period: Overall Study
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev and Anti-PD-1 QW | Arm 2: Lerapolturev and Anti-PD-1 Q3/Q4W
Started | 3 | 12 | 6 | 6
Crossover (Includes participants who started in Arm 1: lerapolturev monotherapy and crossed over to Arm 2: lerapolturev and anti-PD-1) | 1 | 10 | 0 | 0
Completed | 3 | 12 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Lerapolturev QW: lerapolturev weekly for 7 weeks and every 3 weeks thereafter
- Arm 1: Lerapolturev Q3W: lerapolturev at day 1, day 10 and every 3 weeks thereafter includes data from safety run-in
- Arm 2: Lerapolturev + Anti-PD-1 QW: lerapolturev weekly for 7 weeks and every 3 or 4 weeks thereafter anti-PD-1 every 3 or 4 weeks per prescribing information starting at day 1
- Arm 2: Lerapolturev + Anti-PD-1 Q3/4W: lerapolturev at day 1, day 10 and every 3 or 4 weeks thereafter anti-PD-1 every 3 or 4 weeks per prescribing information starting at day 10
- Total: Total of all reporting groups
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W | Total
Number analyzed (Participants) | 3 | 12 | 6 | 6 | 27
Age, Continuous [Mean (Full Range); unit: years] | 60 [44 to 80] | 59 [25 to 84] | 67 [42 to 77] | 65 [53 to 77] | 62 [25 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 4 | 12
  Male | 2 | 8 | 3 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 11 | 5 | 6 | 25
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 12 | 5 | 6 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ECOG Performance Status [Number; unit: patients] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The ECOG Performance Status Scale is a 0-5 point scale where 0 is normal activity with no limitations and 5 is dead. Lower scores indicate a better functional status. A higher score may suggest a poorer prognosis and a greater need for medical care.
  patients
    ECOG PS 0 | 3 | 7 | 2 | 3 | 15
    ECOG PS 1 | 0 | 5 | 4 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: The number of patients achieving confirmed complete (CR) or partial response (PR), per RECIST 1.1 criteria
Time Frame: 24 months
Population: Participants received at least one lerapolturev injection and had at least 1 post-baseline assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 2: Lerapolturev + Anti-PD-1 QW: lerapolturev weekly for 7 weeks and every 3 or 4 weeks thereafter anti-PD-1 every 3 or 4 weeks per prescribing information starting day 1
- Arm 2: Lerapolturev + Anti-PD-1 Q3/4W: lerapolturev at day 1, day 10 and every 3 or 4 weeks thereafter anti-PD-1 every 3 or 4 weeks per prescribing information starting day 10
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
Participants | 0 | 1 | 1 | 0

2. Primary Outcome: Number of Participants Experiencing a Treatment-emergent Adverse Event
Description: The number of participants experiencing a treatment-emergent adverse event
Time Frame: 24 months
Population: The number of participants experiencing a treatment-emergent adverse event are reported here. Detailed data on frequency and severity is reported under Adverse Events.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 6 | 6
Participants | 3 | 10 | 6 | 5

3. Primary Outcome: Number of Participants Experiencing an Adverse Event of Special Interest (AESI) or Anti-PD-1 Immune Related Adverse Events (irAEs)
Description: The number of participants experiencing an AESI or irAE
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 6 | 6
Participants
  Adverse Events of Special Interest | 0 | 0 | 1 | 0
  Immune Related Adverse Events | 0 | 0 | 2 | 0
  No AESI or IrAE reported | 3 | 12 | 3 | 6

4. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to Adverse Event(s)
Description: Number of participants discontinuing study treatment due to adverse event(s)
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 6 | 6
Participants | 0 | 0 | 2 | 1

5. Primary Outcome: Changes From Baseline in the Number of CD8+ Tumor Infiltrating Lymphocytes (TILs)
Description: Changes from baseline in the number of CD8+ tumor infiltrating lymphocytes (TILs)
Time Frame: 24 months
Population: Company ceased operations; samples were not analyzed. Measurement values for this outcome measure are not and will not be available.
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Changes From Baseline in PD-L1 Expression
Description: Changes from baseline in PD-L1 expression
Time Frame: 24 months
Population: as for outcome 5
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS): time from treatment group assignment until death from any cause.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
months | 8.5 [1.5 to NA] — NA = not estimable, insufficient number of participants with events | 4.3 [4.3 to NA] — NA = not estimable, insufficient number of participants with events | NA [9.9 to NA] — NA = not estimable, insufficient number of participants with events | 10.5 [6.3 to NA] — NA = not estimable, insufficient number of participants with events

8. Secondary Outcome: Duration of Response
Description: Duration of Response (DOR): time from confirmed objective response (CR or PR per RECIST 1.1) until unequivocal disease progression or death, whichever occurs first
Time Frame: 24 months
Population: Participants had at least one dose of lerapolturev and at least one post-baseline assessment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
months | NA [NA to NA] — Median and interquartile range are not estimable due to an insufficient number of events; therefore, NA is entered. | NA [NA to NA] — Median and interquartile range are not estimable due to an insufficient number of events; therefore, NA is entered. | NA [NA to NA] — Median and interquartile range are not estimable due to an insufficient number of events; therefore, NA is entered | NA [NA to NA] — Median and interquartile range are not estimable due to an insufficient number of events; therefore, NA is entered

9. Secondary Outcome: Disease Control Rate
Description: The percentage of patients achieving confirmed CR, confirmed PR, or stable disease (SD) per RECIST1.1, as best response.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
percentage of patients | 67 [1 to 91] | 42 [28 to 85] | 60 [5 to 85] | 20 [20 to 99]

10. Secondary Outcome: DCR-6 Months
Description: The number of patients achieving confirmed CR (any duration), confirmed PR (any duration) or SD (≥ 6 months) per RECIST 1.1 as best response.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
Participants | 0 | 1 | 1 | 0

11. Secondary Outcome: Durable Response Rate
Description: The percentage of participants with confirmed CR or PR (per RECIST 1.1) lasting at least 6 months
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
percentage of patients | 0 [0 to 71] | 0 [0 to 26] | 0 [0 to 52] | 0 [0 to 52]

12. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS): time (number of months) from treatment group assignment until date of documented radiologic disease progression per RECIST 1.1 or death due to any cause, whichever comes first
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 3 | 12 | 5 | 5
months | 2.2 [1.3 to NA] — NA = not estimable, insufficient number of participants with events | 1.9 [1.7 to 4.4] | 3.7 [1.4 to NA] — NA = not estimable, insufficient number of participants with events | 1.6 [1.1 to NA] — NA = not estimable, insufficient number of participants with events

13. Other Pre Specified Outcome: Lerapolturev Mechanism of Action and Predictors of Response to Lerapolturev With or Without Anti-PD-1 in Patients Who Have Failed Anti-PD1/L1 -Based Therapy
Description: * Assessment and identification of genetic, cytologic, histologic and/or other markers in tumor biopsies and PBMC samples that may correlate with response.
  * Assessment of changes over time in immune markers, including, but not limited to immune cell density, T cell receptor repertoire, and chemokine and/or cytokine profile in blood, samples, and/or tissue
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: ORR Based on iRECIST
Description: ORR based on iRECIST criteria
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: DOR Based on iRECIST
Description: DOR based on iRECIST criteria
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: DRR Based on iRECIST
Description: DRR based on iRECIST criteria
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: DCR Based on iRECIST
Description: DCR based on iRECIST criteria
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: DCR-6mo Based on iRECIST
Description: DCR-6mo based on iRECIST criteria
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: ORR Based on Subgroup
Description: ORR in the following subgroups:
  * Acquired versus primary PD-1/L1 resistance as defined by Kluger, et al (2020)
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: DOR Based on Subgroup
Description: DOR in the following subgroups:
  * Acquired versus primary PD-1/L1 resistance as defined by Kluger, et al (2020)
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Other Pre Specified Outcome: DRR Based on Subgroup
Description: DRR in the following subgroups:
  * Acquired versus primary PD-1/L1 resistance as defined by Kluger, et al (2020)
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Other Pre Specified Outcome: DCR Based on Subgroup
Description: DCR in the following subgroups:
  * Acquired versus primary PD-1/L1 resistance as defined by Kluger, et al (2020)
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Other Pre Specified Outcome: DCR-6mo Based on Subgroup
Description: DCR-6mo in the following subgroups:
  * Acquired versus primary PD-1/L1 resistance as defined by Kluger, et al (2020)
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Other Pre Specified Outcome: OS Based on Subgroup
Description: OS in the following subgroups:
  * According to treatment arm and AJCC stage at baseline
  * Primary versus acquired resistance as defined by Kluger et al
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Other Pre Specified Outcome: PFS Based on Subgroup
Description: PFS in the following subgroups:
  * According to treatment arm and AJCC stage at baseline
  * Primary versus acquired resistance as defined by Kluger et al
  * BRAF wild type and mutant
  * LDH levels at baseline
  * Time since last dose of anti-PD1/L1 therapy prior to randomization (≤ or >6 weeks)
  * Crossover to combination arm from lerapolturev monotherapy
Time Frame: 24 months
Population: Outcome measure not evaluated
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Arm 1: from treatment start until last dose of study treatment, up to 2 years, or until crossover to Arm 2 Crossover participants: from time of crossover from Arm 1 to Arm 2 until 30 days after last dose of study treatment, up to 2 years Arm 2: from treatment start until last dose of study treatment, up to 2 years
Description: Adverse events were graded using NCI Common Terminology Criteria for Adverse Events v5
Groups:
- Crossover: Initially received lerapolturev (up to 1.6x10^9 TCID50) administered via direct injection. Crossed over to Arm 2: lerapolturev and anti-PD-1. Anti-PD-1 therapy given as per the anti-PD-1 approved package insert.
Arm/Group | Arm 1: Lerapolturev QW | Arm 1: Lerapolturev Q3W | Arm 2: Lerapolturev + Anti-PD-1 QW | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W | Crossover
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/12 | 0/6 | 0/6 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/12 | 2/6 | 2/6 | 3/11
Other Adverse Events (participants affected / at risk) | 3/3 | 10/12 | 6/6 | 5/6 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Lerapolturev QW (N=3) | Arm 1: Lerapolturev Q3W (N=12) | Arm 2: Lerapolturev + Anti-PD-1 QW (N=6) | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W (N=6) | Crossover (N=11)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Lerapolturev QW (N=3) | Arm 1: Lerapolturev Q3W (N=12) | Arm 2: Lerapolturev + Anti-PD-1 QW (N=6) | Arm 2: Lerapolturev + Anti-PD-1 Q3/4W (N=6) | Crossover (N=11)
Fatigue (General disorders) | 1 | 2 | 3 | 0 | 6
Pain (General disorders) | 1 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hypoalbunemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
Blood lactate dehydrogenase increase (Investigations) | 0 | 2 | 0 | 1 | 2
Amylase increased (Investigations) | 1 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 2 | 1 | 1
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT04577807/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04577807/SAP_001.pdf